CLINICAL TRIAL: NCT00004906
Title: A Phase II Multi-Institution Study of Docetaxel and Doxorubicin as Induction Therapy Followed by Sequential High Dose Chemotherapy and CD 34+ Selected Stem Cell Support for Women With Metastatic Breast Cancer
Brief Title: Combination Chemotherapy and Peripheral Stem Cell Transplantation in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NU-H97B1; CDR0000067586 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1682
Record Dates: First submitted 2000-03-07; First posted 2004-08-23 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Filgrastim; Anastrozole; Carboplatin; Cisplatin; Cyclophosphamide; Docetaxel; Doxorubicin; Etoposide; Pamidronate; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: anastrozole
Drug: carboplatin
Drug: cisplatin
Drug: cyclophosphamide
Drug: docetaxel
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: pamidronate disodium
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy plus peripheral stem cell transplantation in treating women who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxicity and response rates to induction therapy with docetaxel and doxorubicin in women with chemotherapy naive metastatic breast cancer. II. Assess the toxicity and response rates to sequential high dose chemotherapy following induction chemotherapy in women with metastatic breast cancer. III. Determine the hematopoietic recovery rate following CD34+ selected peripheral blood stem cell support in this patient population. IV. Assess the toxicity of noncytotoxic maintenance therapy following high dose chemotherapy in this patient population.

OUTLINE: This is a multicenter study. Patients with no prior chemotherapy for metastatic disease receive induction chemotherapy consisting of doxorubicin IV immediately followed by docetaxel IV over 1 hour on day 1. Patients receive filgrastim (G-CSF) subcutaneously (SQ) beginning on day 2 and continuing until day 11-15. Induction therapy repeats every 3 weeks for 4 courses. Within 4 weeks of the last course of induction chemotherapy, patients receive mobilization chemotherapy consisting of cyclophosphamide IV for 2 days, and etoposide IV and cisplatin IV for 3 days. At 24 hours following completion of chemotherapy, patients receive G-CSF SQ twice daily until the target number of peripheral blood stem cells (PBSC) are reached. Within 5 weeks following completion of mobilization chemotherapy, patients receive cyclophosphamide IV, thiotepa IV, and carboplatin IV continuously on days -7 through -4. Patients receive CD34+ selected PBSC on day 0 followed 4 hours later by G-CSF SQ daily and continuing until blood counts recover. Within 30 days of blood count recovery or immediately following completion of post transplantation radiotherapy, patients receive maintenance therapy consisting of oral anastrozole daily until disease progression. Patients with bone involvement also receive pamidronate IV over 2 hours monthly for 1 year. Patients are followed monthly for 6 months, every 3 months for 1 year, every 4-6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed epithelial carcinoma of the breast Metastatic disease including ipsilateral supraclavicular lymph nodes and the chest wall (no axillary nodes) Measurable or evaluable (bone only) disease on exam or radiography No apocrine, adenocystic, squamous cell carcinoma, sarcoma, or lymphoma No symptomatic CNS disease or clinical evidence of CNS metastases Surgically accessible disease Hormone receptor status: Progesterone or estrogen receptor status known

PATIENT CHARACTERISTICS: Age: 18 to 65 Menopausal status: Not specified Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC greater than 3,000/mm3 Platelet count greater than 100,000/mm3 Hepatic: Bilirubin less than 3.0 mg/dL SGOT no greater than 6 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL OR Creatinine clearance greater than 50 mL/min Cardiovascular: Ejection fraction at least 40% by MUGA scan No angina pectoris requiring active nitrate therapy No myocardial infarction within the past 6 months No uncontrolled congestive heart failure No uncontrolled hypertension No major ventricular arrhythmia Other: No uncompensated endocrine dysfunction HIV negative Hepatitis B negative (core antigen negative if vaccinated) No other prior malignancy within the past 5 years except curatively treated nonmelanoma skin cancer or carcinoma in situ of the cervix No active infection or other medical condition that would preclude study Not pregnant Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: At least 6 months since prior adjuvant therapy Biologic therapy: Not specified Chemotherapy: No more than 2 courses of prior induction docetaxel and doxorubicin allowed if staged within 4 weeks of chemotherapy initiation No prior cumulative adjuvant doxorubicin dose greater than 360 mg/m2 No other prior chemotherapy for metastatic disease Endocrine therapy: Prior hormonal therapy for metastatic disease allowed Radiotherapy: Not specified Surgery: See Disease Characteristics

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew L. Pecora, MD, FACP, Study Chair — Hackensack University Medical Center Cancer Center
Locations (4):
- United States (4):
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Ireland Cancer Center, Cleveland, Ohio
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Pecora AL, Lazarus HM, Stadtmauer EA, Winter J, Van Vliet A, Berry D, Gray R, Jennis A, Goldberg S, Cooper BW, Preti R. Effect of induction chemotherapy and tandem cycles of high-dose chemotherapy on outcomes in autologous stem cell transplant for metastatic breast cancer. Bone Marrow Transplant. 2001 Jun;27(12):1245-53. doi: 10.1038/sj.bmt.1703066. PMID 11548842
- [Background] Pecora A, Lazarus H, Stadtmauer E, et al.: Induction chemotherapy prior to sequential high dose chemotherapy compared to no induction increases the rate of complete response and duration of progression free survival in women with metastatic breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 18: A-467, 1999.
- [Result] Pecora AL, Lazarus L, Kramer L, et al.: Phase II multi-institution trial of induction docetaxel and doxorubicin followed by sequential high dose chemotherapy for women with metastatic breast cancer. [Abstract] Proceedings of the American Society of Clinical Oncology 17: A-634, 1998.